CLINICAL TRIAL: NCT06971757
Title: Cost-effectiveness of Routine Follow-up at One Year After Total Hip and Knee Arthroplasty Compared to Check-up on Demand: a Multicenter Hybrid Stepped-wedge Cluster De-implementation Study
Brief Title: HAKA: Routine Follow-Up at 1 Year After Hip- or Knee Arthroplasty: Wasting Resources or Appropriate Healthcare?
Acronym: HAKA 1year FU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JointResearch (Other)
Collaborators: Reinier Haga Orthopedisch Centrum (Other); Tergooi MC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL-009246; 10330042310003 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hip Arthroplasty, Total; Knee Arthroplasty, Total
Keywords: total hip arthroplasty; total knee arthroplasty; follow-up; PROMIS physical function; healthcare consumption

STUDY DESIGN:
Intervention Model Description: This is a hybrid effectiveness (de-)implementation trial type II, with a stepped-wedge cluster trial design. A total of 10 hospitals will transition from a period with RFU to a period with COD, with a wash-out period (transition) of 2 months. The aim is to gradually de-implement RFU, with all centers eventually using COD as the standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Follow-Up (RFU) (Other): X-ray and clinical visit within 3 months and at 1 year after surgery.
  Interventions: Other: Routine Follow-Up (RFU)
- Check-Up on Demand (COD) (Other): X-ray and clinical visit within 3 months and only at 1 year when requested by the patient or healthcare provider.
  Interventions: Other: Check-Up on Demand (COD)

INTERVENTIONS:
Other: Routine Follow-Up (RFU) — Standard follow-up care with scheduled X-ray and clinical visit at 3 months and 1 year after surgery.
  Arms: Routine Follow-Up (RFU)
Other: Check-Up on Demand (COD) — Follow-up care with scheduled X-ray and clinical visit at 3 months and only at 1 year if requested.
  Arms: Check-Up on Demand (COD)

SUMMARY:
After undergoing total hip or total knee arthroplasty, current guidelines recommend routine follow-up with an X-ray within 3 months and again at 1 year. Follow-up at 5 years (for hip arthroplasties) or every 5 years (for knee arthroplasties) is also considered worthwhile according to the guideline. However, these follow-up appointments require considerable time from patients, caregivers, and healthcare professionals, and it is unclear whether they are truly beneficial. It is possible that a single follow-up within 3 months is sufficient. This could potentially prevent over 100,000 unnecessary hospital visits per year, resulting in significant cost savings. If patients or healthcare providers have concerns, they can always request an additional follow-up.

The HAKA trial consists of three different work packages (WPs). This trial (WP1) investigates the 1-year follow-up, WP2 examines the 10-year follow-up, and WP3 is a qualitative study exploring the experiences and perceptions of patients and healthcare professionals. The aim of the HAKA trial is to safely reduce routine follow-up appointments after total hip or knee arthroplasty and to revise current clinical guidelines accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Painful and disabled hip or knee joint resulting from osteoarthritis
* Scheduled for primary THA or TKA surgery
* Age 50 years or older at the time of THA or TKA
* Capable and willing to complete questionnaires
* Proficient in Dutch or English
* Willing to provide informed consent

Exclusion Criteria:

* Other indication for surgery than osteoarthritis
* Scheduled for hip or knee revision arthroplasty, except a conversion from unicompartmental knee arthroplasty to TKA or from hip hemiarthroplasty/resurfacing to THA
* Already participating in this study due to a previous hip or knee surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS Physical Function | Assessed before surgery and at 3, 12, 15, 18, and 24 months after surgery.
  Patient-reported physical functioning will be assessed using the PROMIS® Physical Function Version 1.0, Short Form 10a. The short form consists of 10 items and is expressed by raw summed score ranging from 10 to 50, which can be converted to a T-score and SE. The T-score is a standardized score with a mean of 50 and a SD of 10. Higher T-scores indicate better physical functioning.
Number of clinical visits and X-rays | From surgery until 24 months after surgery.
  Assesses healthcare consumption based on the number of postoperative outpatient clinical visits and X-ray assessments.

SECONDARY OUTCOMES:
Number of complications | From surgery until 24 months after surgery.
  The total number of post-operative complications per patient will be recorded.
Type of Complications | From surgery until 24 months after surgery.
  Complication types will be recorded and categorized (e.g., infection, periprosthetic fracture, loosening, malalignment, dislocation, prosthetic wear).
Number of surgical interventions | From surgery until 24 months after surgery.
  The total number of surgical re-interventions per patient related to the index procedure will be recorded.
Type of Surgical Interventions | From surgery until 24 months after surgery
  Types of surgical re-interventions will be recorded and categorized (e.g., DAIR, partial component exchange, full revision, irrigation and debridement without component retention).
Costs related to THA or TKA follow-up | Assessed at 15, 18, and 24 months after surgery.
  Includes costs from electronic health records and additional patient questionnaires, covering hospital and non-hospital care.
Numeric Pain Rating Scale (NPRS) | Assessed before surgery and at 3, 12, 15, 18, and 24 months after surgery.
  Patient-reported pain intensity, measured using a numeric scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores reflect more severe pain.
EQ-5D-5L | Assessed before surgery and at 3, 12, 15, 18, and 24 months after surgery.
  Health-related quality of life is measured using the EQ-5D-5L questionnaire. The EQ-5D-5L index score ranges from -0.594 to 1.000, where 1.000 indicates full health, 0 represents death, and negative values represent health states worse than death. Higher scores indicate better health status.

CONTACTS AND LOCATIONS:
Locations (9):
- Netherlands (9):
  - OLVG, Amsterdam
  - Amphia, Breda
  - Deventer Ziekenhuis, Deventer
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Martini Ziekenhuis, Groningen
  - Tergooi MC, Hilversum
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - ZorgSaam Zeeuws Vlaanderen, Terneuzen
  - RHOC, Zoetermeer

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in publications (e.g., PROMs, healthcare consumption, complications) will be made available upon reasonable request. Metadata will be openly accessible with a persistent identifier.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available beginning 6 months after publication of the main results and will remain available for at least 5 years thereafter.
Access Criteria: Researchers who provide a methodologically sound proposal and agree to a data use agreement will be granted access to de-identified IPD and selected supporting documents. Requests can be submitted to the corresponding author or data access contact. Access is conditional on approval by the study team.

REFERENCES:
- See also: Related Info — https://zorgevaluatienederland.nl/evaluations/haka-1-year-fu